CLINICAL TRIAL: NCT03789292
Title: A Randomized, Active-Controlled, Double-Blind, Phase 3 Study to Compare Efficacy and Safety of CT-P17 With Humira When Co-administered With Methotrexate in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: A Study to Compare Efficacy and Safety of CT-P17 With Humira in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P17 3.1; 2018-001690-25 (EudraCT Number)
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-P17 Subcutaneous(SC) (adalimumab) (Experimental): CT-P17 SC (adalimumab)
  Interventions: Biological: CT-P17 SC
- Humira SC (adalimumab) (Active Comparator): Humira SC (adalimumab)
  Interventions: Biological: CT-P17 SC; Biological: Humira SC

INTERVENTIONS:
Biological: CT-P17 SC — Subcutaneous injection of Adalimumab 40mg every two weeks
Biological: Humira SC — Subcutaneous injection of Adalimumab 40mg every two weeks
  Arms: Humira SC (adalimumab)

SUMMARY:
This is a Phase III Study to Compare Efficacy and Safety of CT-P17 with Humira in Patients With Active Rheumatoid Arthritis

DETAILED DESCRIPTION:
CT-P17, containing the active ingredient adalimumab, is a recombinant humanized monoclonal antibody that is being developed as a similar biological medicinal product to Humira. The purpose of this study is to demonstrate similar efficacy and safety of CT-P17 and Humira in patients with moderate to severe rheumatoid arthritis when co-administered with methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female aged 18 to 75 years old, both inclusive.
* Patient has had a diagnosis of rheumatoid arthritis according to the 2010 American College of Rheumatology(ACR)/EULAR classification criteria for at least 24 weeks prior to the first administration of the study drug .

Exclusion Criteria:

* Patient who has previously received investigational or licensed product; biologic or targeted synthetic disease-modifying antirheumatic drugs for the treatment of rheumatoid arthritis and/or a tumor necrosis factor (TNF) α inhibitor for any purposes.
* Patient who has allergies to any of the excipients of study drug or any other murine and human proteins, or patient with a hypersensitivity to immunoglobulin products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MinJi Ma, Study Chair — Celltrion, Inc.
Locations (1):
- National Multiprofile Transport Hospital Tsar Boris III, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furst DE, Jaworski J, Wojciechowski R, Wiland P, Dudek A, Krogulec M, Jeka S, Zielinska A, Trefler J, Bartnicka-Maslowska K, Krajewska-Wlodarczyk M, Klimiuk PA, Lee SJ, Kim SH, Bae YJ, Yang GE, Yoo JK, Kay J, Keystone E. Efficacy and safety of switching from reference adalimumab to CT-P17 (100 mg/ml): 52-week randomized, double-blind study in rheumatoid arthritis. Rheumatology (Oxford). 2022 Apr 11;61(4):1385-1395. doi: 10.1093/rheumatology/keab460. PMID 34142111
- [Derived] Kay J, Jaworski J, Wojciechowski R, Wiland P, Dudek A, Krogulec M, Jeka S, Zielinska A, Trefler J, Bartnicka-Maslowska K, Krajewska-Wlodarczyk M, Klimiuk PA, Lee SJ, Bae YJ, Yang GE, Yoo JK, Furst DE, Keystone E. Efficacy and safety of biosimilar CT-P17 versus reference adalimumab in subjects with rheumatoid arthritis: 24-week results from a randomized study. Arthritis Res Ther. 2021 Feb 5;23(1):51. doi: 10.1186/s13075-020-02394-7. PMID 33546755

RESULTS

PARTICIPANT FLOW:
Groups:
- CT-P17 Subcutaneous(SC) (Adalimumab): Treatment Period 1: On Day 1 (Week 0), patients were randomly assigned to receive either CT-P17 or EU-approved Humira (40mg/0.4mL each) administered by subcutaneous (SC) injection via pre-filled syringe (PFS) every other week (EOW) in combination with methotrexate (MTX) and folic acid from Week 0 to Week 24.
  Treatment Period 2: All patients who were initially randomly assigned to CT-P17 (40mg/0.4mL) at Day 1 (Week 0) continued their treatment with CT-P17 from Week 26 up to Week 48.
- EU-approved Humira SC (Adalimumab): Treatment Period 1: On Day 1 (Week 0), patients were randomly assigned to receive either CT-P17 or EU-approved Humira (40mg/0.4mL each) administered by subcutaneous (SC) injection via pre-filled syringe (PFS) every other week (EOW) in combination with methotrexate (MTX) and folic acid from Week 0 to Week 24.
  Treatment Period 2: Patients who were initially randomly assigned to EU-approved Humira were randomized again prior dosing at Week 26, in a ratio of 1:1 to either continue EU-approved Humira or undergo transition to CT-P17 (40mg/0.4mL each) from Week 26 to Week 48.
- Switched to CT-P17: Treatment Period 1: N/A
  Treatment Period 2: Patients who were initially randomly assigned to EU-approved Humira were randomized again prior dosing at Week 26, in a ratio of 1:1 to either continue EU-approved Humira or undergo transition to CT-P17 (40mg/0.4mL each) from Week 26 to Week 48.
Period: Treatment Period I (Week 0 to Week 26)
Arm/Group | CT-P17 Subcutaneous(SC) (Adalimumab) | EU-approved Humira SC (Adalimumab) | Switched to CT-P17
Started | 324 | 324 | 0
Completed | 303 | 305 | 0
Not Completed | 21 | 19 | 0
Not completed — Adverse Event | 7 | 8 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 9 | 8 | 0
Not completed — Significant dose delay | 1 | 0 | 0
Not completed — Patient decision | 0 | 2 | 0
Period: Treatment Period II (Week 26 to Week 52)
Arm/Group | CT-P17 Subcutaneous(SC) (Adalimumab) | EU-approved Humira SC (Adalimumab) | Switched to CT-P17
Started | 303 | 153 (Patients who had administrated Humira SC during Treatment Period 1 has been devided into 2 groups - maintaining Humira SC and switched to CT-P17.) | 152 (Patients who had administrated Humira SC during Treatment Period 1 has been devided into 2 groups - maintaining Humira SC and switched to CT-P17.)
Completed | 287 | 147 | 143
Not Completed | 16 | 6 | 9
Not completed — Adverse Event | 3 | 3 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 2 | 2
Not completed — Significant dose delay | 1 | 0 | 0
Not completed — Could not visit the site due to COVID-19 pandemic | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CT-P17: Patients were administered CT-P17 (40mg/0.4mL) by SC injection via PFS EOW in combination with MTX and folic acid from Week 0 to Week 24.
- EU-approved Humira: Patients were administered EU-approved Humira (40mg/0.4mL) by SC injection via PFS EOW in combination with MTX and folic acid from Week 0 to Week 24.
- Total: Total of all reporting groups
Arm/Group | CT-P17 | EU-approved Humira | Total
Number analyzed (Participants) | 324 | 324 | 648
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 268 | 282 | 550
  >=65 years | 55 | 42 | 97
Age, Continuous [Median (Full Range); unit: years] | 53.5 [18 to 75] | 54.0 [19 to 75] | 54.0 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249 | 265 | 514
  Male | 75 | 59 | 134
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 299 | 298 | 597
  Race: Other | 25 | 26 | 51
Region of Enrollment [Count of Participants; unit: Participants]
  Bulgaria | 20 | 19 | 39
  Hungary | 17 | 17 | 34
  Lithuania | 4 | 5 | 9
  Peru | 25 | 26 | 51
  Poland | 231 | 231 | 462
  Ukraine | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology(ACR)20 Response Rate at Week 24.
Description: ACR20 is defined as both improvement of 20% in the number of tender and number of swollen joints, and a 20% improvement in the three of the following five criteria: 1) patient global assessment of disease activity, 2) physician global assessment of disease activity, 3) functional ability measure using Health Assessment Questionnaire (HAQ), 4) visual analog pain scale, and 5) erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)
Time Frame: Week 24
Population: Intent-to-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P17 Subcutaneous(SC) (Adalimumab) | EU-approved Humira SC (Adalimumab)
Number analyzed (Participants) | 324 | 324
Participants | 268 | 268

2. Secondary Outcome: ACR50 and ACR70 Response Rate at Week 24
Description: ACR50 and ACR70 are the same instruments with improvement levels defined as 50% and 70% respectively versus 20% for ACR20.
Time Frame: Week 24
Population: Intent-to-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P17 | EU-approved Humira
Number analyzed (Participants) | 324 | 324
Participants
  ACR50 at Week 24 | 195 | 206
  ACR70 at Week 24 | 132 | 144

3. Secondary Outcome: ACR20, ACR50, and ACR70 Response Rate up to Week 52
Description: ACR20 is defined as both improvement of 20% in the number of tender and number of swollen joints, and a 20% improvement in the three of the following five criteria: 1) patient global assessment of disease activity, 2) physician global assessment of disease activity, 3) functional ability measure using Health Assessment Questionnaire (HAQ), 4) visual analog pain scale, and 5) erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP). ACR50 and ACR70 are the same instruments with improvement levels defined as 50% and 70% respectively versus 20% for ACR20.
Time Frame: Up to Week 52
Population: Intent-to-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Groups:
- CT-P17 Maintenance: All patients who were initially randomly assigned to CT-P17 (40mg/0.4mL) at Day 1 (Week 0) continued their treatment with CT-P17 from Week 26 up to Week 48.
- Humira Maintenance; Switched to CT-P17: Patients who were initially randomly assigned to EU-approved Humira were randomized again prior dosing at Week 26, in a ratio of 1:1 to either continue EU-approved Humira or undergo transition to CT-P17 (40mg/0.4mL each) from Week 26 to Week 48.
Arm/Group | CT-P17 Maintenance | Humira Maintenance | Switched to CT-P17
Number analyzed (Participants) | 303 | 153 | 152
Participants
  ACR20 at Week 52 | 244 | 119 | 125
  ACR50 at Week 52 | 201 | 95 | 101
  ACR70 at Week 52 | 135 | 75 | 72

4. Secondary Outcome: Mean Change From Baseline in Disease Activity Measured by DAS28 (CRP)
Description: The Disease activity score (DAS28) (c-reactive protein [CRP]) score was derived using the following formulae:
  DAS28 (CRP) = 0.56*√(TJC28) + 0.28*√(SJC28) + 0.014*(GH) + 0.36*ln(CRP+1) + 0.96
  Where:
  TJC28 = 28 joint count for tenderness (0-28) SJC28 = 28 joint count for swelling (0-28) Ln (CRP) = natural logarithm of CRP (mg/L : 0.2-236.3 as observed in the study) GH = General Health component of the DAS (patient's global assessment of disease activity) (mm: 0-100).
  DAS28 (CRP) values range from 1.03 to 8.77 while higher values mean a higher disease activity.
Time Frame: Week 24
Population: Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CT-P17 | EU-approved Humira
Number analyzed (Participants) | 324 | 324
Units on a scale | -2.738 (1.1911) | -2.734 (1.2052)

5. Secondary Outcome: Mean Change From Baseline in Disease Activity Measured by DAS28 (CRP)
Description: as for outcome 4
Time Frame: Up to Week 52
Population: Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CT-P17 Maintenance | Humira Maintenance | Switched to CT-P17
Number analyzed (Participants) | 303 | 153 | 152
Units on a scale | -2.945 (1.1273) | -3.074 (1.1926) | -2.983 (1.2529)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the date the patient signed the Informed Consent Form(ICF) until 4 weeks after the last study drug administration (up to 52 weeks).
Description: Treatment Period I: Week 0 to Week 26 pre-dose Treatment Period II: Week 26 to Week 52 end of study visit
Groups:
- Treatment 1: CT-P17: Patients were administered CT-P17 (40mg/0.4mL) by SC injection via PFS EOW in combination with MTX and folic acid from Week 0 to Week 24.
- Treatment 1: EU-approved Humira: Patients were administered EU-approved Humira (40mg/0.4mL) by SC injection via PFS EOW in combination with MTX and folic acid from Week 0 to Week 24.
- Treatment 2: CT-P17 Maintenance: All patients who were initially randomly assigned to CT-P17 (40mg/0.4mL) at Day 1 (Week 0) continued their treatment with CT-P17 from Week 26 up to Week 48.
- Treatment 2: Humira Maintenance; Treatment 2: Switched to CT-P17: Patients who were initially randomly assigned to EU-approved Humira were randomized again prior dosing at Week 26, to either continue EU-approved Humira or undergo transition to CT-P17 (40mg/0.4mL each) from Week 26 to Week 48.
Arm/Group | Treatment 1: CT-P17 | Treatment 1: EU-approved Humira | Treatment 2: CT-P17 Maintenance | Treatment 2: Humira Maintenance | Treatment 2: Switched to CT-P17
All-Cause Mortality (participants affected / at risk) | 0/324 | 0/324 | 0/303 | 0/152 | 0/152
Serious Adverse Events (participants affected / at risk) | 12/324 | 19/324 | 6/303 | 3/152 | 5/152
Other Adverse Events (participants affected / at risk) | 96/324 | 118/324 | 50/303 | 35/152 | 33/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1: CT-P17 (N=324) | Treatment 1: EU-approved Humira (N=324) | Treatment 2: CT-P17 Maintenance (N=303) | Treatment 2: Humira Maintenance (N=152) | Treatment 2: Switched to CT-P17 (N=152)
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vitreous hemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Extradural hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Benign muscle neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Ischemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Cataract operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Polypectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1: CT-P17 (N=324) | Treatment 1: EU-approved Humira (N=324) | Treatment 2: CT-P17 Maintenance (N=303) | Treatment 2: Humira Maintenance (N=152) | Treatment 2: Switched to CT-P17 (N=152)
Leukopenia (Blood and lymphatic system disorders) | 10 | 9 | 8 | 0 | 7
Neutropenia (Blood and lymphatic system disorders) | 13 | 17 | 15 | 6 | 8
Diarrhea (Gastrointestinal disorders) | 5 | 3 | 2 | 3 | 5
Injection site reaction (General disorders) | 16 | 23 | 1 | 4 | 1
Latent tuberculosis (Infections and infestations) | 12 | 15 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 17 | 20 | 6 | 5 | 3
Pharyngitis (Infections and infestations) | 12 | 10 | 4 | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 18 | 22 | 10 | 11 | 6
Urinary tract infection (Infections and infestations) | 15 | 15 | 9 | 5 | 3
Alanine aminotransferase increased (Investigations) | 11 | 17 | 8 | 1 | 7
Aspartate aminotransferase increased (Investigations) | 4 | 12 | 4 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT03789292/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT03789292/SAP_001.pdf